CLINICAL TRIAL: NCT02926053
Title: T Cell Therapy for Patients With Metastatic Renal Cell Carcinoma
Brief Title: TIL Therapy for Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, MD, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UG1617
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient group (Experimental): All patients receive the same treatment.
  Surgical removal of tumor tissue for T cell production, which takes 4-6 weeks, is performed initially.
  All patients are hospitalized during treatment (one week in advance of the T cell product being ready and for approximately 3 weeks in total) and receive treatment only once.
  The patients are admitted to hospital day -8 and receive lymphodepleting chemotherapy (cyclophosphamide and fludarabine on day -7 to day -1.
  The TILs are infused on day 0 and Interleukin-2 therapy is administered on day 0 to day 5. Interleukin-2 is administered as high-dose i.v. bolus every eight hour starting approximately 6 hours after TIL infusion and for up to 5 days (maximum of 15 doses).
  Interventions: Procedure: Surgical removal of tumor tissue for T cell production; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: TIL infusion; Drug: Interleukin-2

INTERVENTIONS:
Procedure: Surgical removal of tumor tissue for T cell production — Surgical removal of > 1 cm3 tumor tissue chosen with regards to high rate of success and to minimize the general risks involved in a surgical procedure.
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg is administered i.v. on day -7 and day -6.
  Other Names: Cyclophospamide
Drug: Fludarabine — Fludarabine 25 mg/m2 is administered on day -5 to day -1. Maximum dose of 50 mg per administration.
  Other Names: Fludarabinephosphate; Fludara
Biological: TIL infusion — The maximum number of expanded TILs are infused over 30-45 minutes on day 0.
  Other Names: T Cell infusion
Drug: Interleukin-2 — Interleukin-2 is administered as high-dose bolus infusions (600.000 IU/kg) over a 15 minute period every 8 hours and continuing for up to 5 days (maximum of 15 doses).
  Other Names: IL-2; Proleukin

SUMMARY:
Adoptive T cell therapy (ACT) with tumor infiltrating lymphocytes (TIL) has achieved impressive clinical results with durable complete responses in patients with metastatic melanoma. The TILs are isolated from patients own tumor tissue followed by in vitro expansion and activation for around 4-6 weeks. Before TIL infusion the patients receive 1 week of preconditioning chemotherapy with cyclophosphamide and fludarabine. After TIL infusion Interleukin-2 is administered to support T cell activation and proliferation in vivo.

Recent studies suggest, that TIL therapy works in other cancers than Metastatic Melanoma, including Renal Cell Carcinoma. In this study TIL therapy is administered to patients with metastatic Renal Cell Carcinoma.

DETAILED DESCRIPTION:
Adoptive T cell therapy (ACT) with tumor infiltrating lymphocytes (TIL) has achieved impressive clinical results with durable complete responses in patients with metastatic melanoma. The TILs are isolated from patients own tumor tissue followed by in vitro expansion and activation for around 4-6 weeks. Before TIL infusion the patients receive 1 week of preconditioning chemotherapy with cyclophosphamide and fludarabine. After TIL infusion Interleukin-2 is administered to support T cell activation and proliferation in vivo.

Objectives:

To evaluate safety and feasibility when treating patients with metastatic renal cell carcinoma with ACT with TILs.

To evaluate treatment related immune responses . To evaluate clinical efficacy.

Design:

Patients will be screened with a physical exam, medical history, blood samples, pulmonary function test, Cr-EDTA clearance, MUGA scan and ECG.

Patients will undergo surgery to harvest tumor material for TIL production.

Patients is admitted day -8 in order to undergo lymphodepleting chemotherapy with cyclophosphamide and fludara starting day -7.

On day 0 patients receive TIL infusion and shortly after starts IL-2 administration with high-dose bolus IL-2 every eight hour for up to 5 days (maximum of 15 doses).

The patients will followed until progression or up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven mRCC with the possibility of surgical removal of tumor tissue of > 1 cm3. Histology must include a clear cell component with or without a sarcomatoid dedifferentiation.
* Metastatic disease irrespective of number of previous treatment lines. Treatment naïve pt's can be included.
* ECOG performance status of ≤1.
* IMDC prognostic group 'Favorable' or 'Intermediary'.
* Life expectancy of > 6 months.
* At least one measurable parameter after surgery in accordance with RECIST 1.1 -criteria's.
* No significant toxicities or side effects (CTC ≤ 1) from previous treatments.
* Normal ejection fraction (EF) measured by a multigated acquisition (MUGA) scan.
* Crom EDTA clearance >40 ml/min.
* Adequate renal, hepatic and hematological function.
* LDH ≤ 5 times upper normal limit as a measure of tumor burden.
* Women in the fertile age must use effective contraception. Likewise, men included in the study, as well as their partners, must use effective contraception. This applies from inclusion and until 6 months after treatment. Birth control pills, spiral, depot injection with gestagen, subdermal implantation, hormonal vaginal ring and transdermal depot patch are all considered safe contraceptives.
* Able to comprehend the information given and willing to sign informed consent.
* Willingness to participate in the planned controls.

Exclusion Criteria:

* A history of prior malignancies, except curatively treated non-melanoma skin cancer and CIS of the cervix uteri. Patients treated for another malignancy can participate if they are without signs of disease for a minimum of 3 years after treatment.
* Patients with cerebral metastases.
* Patients with widespread bone or bone only metastases.
* Severe allergies, history of anaphylaxis or known allergies to the administered drugs.
* Severe medical conditions or psychiatric comorbidity.
* Acute/chronic infection with HIV, hepatitis, tuberculosis among others.
* Severe and active autoimmune disease.
* Pregnant women and women breastfeeding.
* Simultaneous treatment with systemic immunosuppressive drugs (including prednisolone, methotrexate among others).
* Simultaneous treatment with other experimental drugs.
* Simultaneous treatment with other systemic anti-cancer treatments.
* Patients with active and uncontrollable hypercalcaemia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-12; Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inge M Svane, Prof., MD, Study Director — Center for Cancer Immune Therapy, Department of Oncology, Herlev Hospital, Borgmester Ib Juuls vej 25C, DK-2730; Troels H Borch, MD, PhD, Principal Investigator — Center for Cancer Immune Therapy, Department of Oncology, Herlev Hospital, Borgmester Ib Juuls vej 25C, DK-2730
Locations (1):
- Center for Cancer Immune Therapy Dept. of Hematology/oncology, Herlev, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Group: All patients receive the same treatment.
  Surgical removal of tumor tissue for T cell production, which takes 4-6 weeks, is performed initially.
  All patients are hospitalized during treatment (one week in advance of the T cell product being ready and for approximately 3 weeks in total) and receive treatment only once.
  The patients are admitted to hospital day -8 and receive lymphodepleting chemotherapy (cyclophosphamide and fludarabine on day -7 to day -1.
  The TILs are infused on day 0 and Interleukin-2 therapy is administered on day 0 to day 5. Interleukin-2 is administered as high-dose i.v. bolus every eight hour starting approximately 6 hours after TIL infusion and for up to 5 days (maximum of 15 doses).
  Surgical removal of tumor tissue for T cell production: Surgical removal of > 1 cm3 tumor tissue chosen with regards to high rate of success and to minimize the general risks involved in a surgical procedure.
  Cyclophosphamide: Cyclophosphamide 60 mg/kg is administered i.v. on day -7 and day -6.
  Fludarabine: Fludarabine 25 mg/m2 is administered on day -5 to day -1. Maximum dose of 50 mg per administration.
  TIL infusion: The maximum number of expanded TILs are infused over 30-45 minutes on day 0.
  Interleukin-2: Interleukin-2 is administered as high-dose bolus infusions (600.000 IU/kg) over a 15 minute period every 8 hours and continuing for up to 5 days (maximum of 15 doses).
Period: Overall Study
Arm/Group | Patient Group
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patient Group
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Which the Treatment Was Tolerable
Description: Determine the safety of the administration of TIL therapy including lymphodepleting chemotherapy and Interleukin-2 for patients with metastatic renal cell cancer. This will be assessed clinically by whether the patients are able to receive treatment as described in the protocol.
Time Frame: 0-24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Group
Number analyzed (Participants) | 5
Participants | 5

2. Secondary Outcome: Number of Infusion Products With Detectable in Vitro Anti-tumor Responses
Description: In vitro anti-tumor responses will be measured by cytokine production in a flow-cytometry based assed after co-culture of tumor-infiltrating lymphocytes from the infusion product with autologous tumor cells (from tumor digest and/or autologous tumor cell lines).
Time Frame: Up to 12 months
Measure: Number; unit: Infusion products
Arm/Group | Patient Group
Number analyzed (Participants) | 5
Infusion products | 4

3. Secondary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Group
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected continuously during the trial from inclusion to end-of-study visit, up to 9 months.
Arm/Group | Patient Group
All-Cause Mortality (participants affected / at risk) | 4/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Group (N=5)
Hypotension (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient Group (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Petechiae (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 5
Dyspnoe (Respiratory, thoracic and mediastinal disorders) | 5
Confusional state (Nervous system disorders) | 2
Hallucination (Nervous system disorders) | 1
Fatigue (General disorders) | 5
Pain (General disorders) | 4
Performance status decreased (General disorders) | 5
Weight increased (General disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Melaena (Gastrointestinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Infection (Infections and infestations) | 4

LIMITATIONS AND CAVEATS:
The trial was designed to include six patients, but due to very slow recruitment the trial only included five patients which is an obvious limitation of the trial and limits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT02926053/Prot_000.pdf